CLINICAL TRIAL: NCT07060560
Title: Prospective Observational Study to Evaluate the Diagnostic Accuracy of Presepsin for Sepsis in Severe Burn Patients
Brief Title: Presepsin Diagnostic Performance in Severe Burn Sepsis
Acronym: PSEP-BURNS
Status: Recruiting | Type: Observational
Sponsor: Dohern Kym (Other)
Responsible Party: Sponsor-Investigator, Dohern Kym, Attending Physician, Burn Intensive Care Unit, Hangang Sacred Heart Hospital
Organization: Hangang Sacred Heart Hospital (Other)
Other Study IDs: 2025-009
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Sepsis; Burns
MeSH Terms: conditions — Sepsis; Burns

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Days
Oversight: Data Monitoring Committee: No

SUMMARY:
This study enrolls approximately 270 adult patients with severe burns covering at least 20% of total body surface area to evaluate how well the blood biomarker presepsin diagnoses sepsis early in this high-risk population. Sepsis-a life-threatening condition caused by an exaggerated immune response to infection-is particularly urgent to detect promptly in burn patients. Participants will undergo blood tests for presepsin at predefined time points, and these results will be compared to C-reactive protein (CRP), procalcitonin (PCT) levels, Sepsis-3 clinical criteria, and blood culture findings. The primary goal is to measure presepsin's sensitivity and specificity for sepsis detection, thereby determining its diagnostic accuracy. Findings from this study may enable faster sepsis treatment in severe burn patients and improve clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 18 years admitted to Hangang Sacred Heart Hospital Burn ICU with total body surface area (TBSA) ≥ 20 %
* Clinical suspicion of sepsis prompting blood culture and biomarker sampling
* Ability to understand the study and provide written informed consent (or via legally authorized representative)

Exclusion Criteria:

* Inability to undergo research blood draw due to emergent surgery or major trauma at sampling time
* Chronic immunosuppressive conditions (e.g., long-term high-dose steroids, organ transplant, congenital immunodeficiency)
* Pregnant women or those with significant psychiatric conditions precluding consent
* Any other medical or safety concerns deemed inappropriate by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A prospective cohort of adult (≥ 18 years) patients with severe burns (TBSA ≥ 20 %) admitted to the Burn Intensive Care Unit at Hangang Sacred Heart Hospital
Sampling Method: Non-Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic sensitivity and specificity of presepsin for sepsis in severe burn patients | Up to 2 hours after initial clinical suspicion of sepsis.
  The proportion of true-positive and true-negative presepsin results for diagnosing sepsis using Sepsis-3 clinical criteria and positive blood culture as the reference standard.

CONTACTS AND LOCATIONS:
Locations (1):
- Hangang Sacred Heart Hospital, Hallym University Medical Center, Seoul, Seoul, South Korea